CLINICAL TRIAL: NCT07297329
Title: A Phase 3 Randomized, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of SCTC21C in Combination With Bortezomib, Lenalidomide and Dexamethasone Versus Bortezomib, Lenalidomide and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Not Eligible for Transplant
Brief Title: A Study to Evaluate the Safety and Efficacy of SCTC21C in Combination With Bortezomib, Lenalidomide and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Not Eligible for Transplant
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCTC21C-A301
Record Dates: First submitted 2025-12-03; First posted 2025-12-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCTC21C + VRd (S-VRd) (Experimental)
  Interventions: Drug: SCTC21C; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- VRd (Active Comparator)
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: SCTC21C — Pharmaceutical form: Solution for infusion； Route of administration: Subcutaneous
  Arms: SCTC21C + VRd (S-VRd)
Drug: Bortezomib — Pharmaceutical form: Lyophilized powder for injection； Route of administration: Subcutaneous
Drug: Lenalidomide — Pharmaceutical form: Capsules； Route of administration: Oral
Drug: Dexamethasone — Pharmaceutical form: Tablets, ampoules or vials for injection； Route of administration: Oral/Intravenous

SUMMARY:
The purpose of this study is to evaluate if the addition of SCTC21C to bortezomib, lenalidomide and dexamethasone (VRd) in patients with newly diagnosed multiple myeloma not eligible for transplant will prolong progression-free survival (PFS) and/or improve overall minimal residual disease (MRD) negativity rate compared with VRd alone.

DETAILED DESCRIPTION:
This study comprises two phases: Part 1 is the safety run in, while Part 2 is a randomized, controlled, open-label, multicenter study. Both parts are divided into three stages: the screening period (up to 28 days before first dose/randomization), the treatment period (from Cycle 1 [28 days] Day 1 and continues until disease progression or unacceptable toxicity), and the follow-up period (Postintervention). Safety endpoints include treatment-emergent adverse events , treatment-related adverse events, serious adverse events, clinical laboratory tests, vital signs, physical examinations, electrocardiograms , etc. Efficacy endpoints include objective response rate (ORR), progression-free survival (PFS), and minimal residual disease (MRD) negativity rate.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed multiple myeloma (IMWG criteria) not eligible for transplant.
* Evidence of measurable disease.
* With adequate organ function and hematological parameters.
* Contraception，and during the study period and for 5 months after the last dose, all subjects must not donate reproductive cells.

Exclusion Criteria:

* Other hematologic malignancies.
* Subjects with confirmed or suspected central nervous system infiltration or meningeal involvement.
* Uncontrolled infection.
* Subjects with conditions that may affect safety or efficacy assessments include, but are not limited to, cardiovascular, respiratory, endocrine/metabolic, immune system, hepatic, gastrointestinal (such as gastrointestinal bleeding, perforation, ulcers, etc.), and malignant neoplasms, and are deemed clinically significant by the investigator.
* Subjects who have undergone major surgery or experienced significant trauma within 4 weeks prior to the first use of the investigational drug, or who require elective surgery during the trial period.
* Received a live or attenuated vaccine within 30 days prior to the first dose; Female subjects who are currently breastfeeding.
* Subjects with mental disorders or poor compliance, or other circumstances deemed unsuitable for participation in this study by other investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 84 months after the First Participant In (FPI)
  Defined as the time from the date of randomization to the date of first documentation of progression disease (PD) or the date of death from any cause, whichever occurs first.
Minimal residual disease (MRD) negativity rate for participants with CR | Up to approximately 84 months after the FPI
  Proportion of participants with CR for whom MRD measurement is negative

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 84 months after the FPI
  Proportion of participants with best overall response (BOR) recorded as sCR, CR, VGPR, or partial response (PR) using the IMWG criteria
Duration of response (DOR) | Up to approximately 84 months after the FPI
  Defined as the time from date of first response to date of first PD or death, whichever occurs first for participants achieving sCR, CR, VGPR, or PR
Adverse Events | Up to approximately 84 months after the FPI
  Treatment-emergent adverse events/serious adverse events

OTHER OUTCOMES:
PRO: EQ-5D-5L | Up to approximately 84 months after the FPI
  Health state utility and health status will be assessed using the European Quality of Life Group questionnaire with 5 dimensions and 5 levels per dimension (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China